CLINICAL TRIAL: NCT00633815
Title: Study of Upright Versus Supine Exercise Testing in Fontan-palliated Patients, Compared With Healthy Controls, to Evaluate for Postural Effects on Exercise Parameters
Brief Title: Upright Versus Supine Exercise Testing in Fontan-palliated Patients
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Bryan Goldstein, Fellow, Pediatric Cardiology, University of Michigan
Other Study IDs: HUM00007190
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Fontan Palliation
Keywords: Supine; Upright
MeSH Terms: conditions — Deception

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fontan patients: Subjects will undergo exercise testing in both the supine and upright positions
  Interventions: Other: Supine positioning; Other: Upright positioning
- Healthy controls: Subjects will undergo exercise testing in both the supine and upright positions
  Interventions: Other: Supine positioning; Other: Upright positioning

INTERVENTIONS:
Other: Supine positioning — Subjects underwent exercise testing on a stationary bicycle in the supine position
Other: Upright positioning — Subjects underwent exercise testing on a stationary bicycle in the upright position

SUMMARY:
Fontan-palliated patients comprise an interesting group of single-ventricle patients who are dependent upon passive return of blood from the body to the lungs. Systemic venous pressures are therefore quite elevated, and one study demonstrated that venous capacitance was diminished. In addition, these patients have markedly diminished aerobic capacity (Max VO2). Although one recent study demonstrated that Fontan patients can increase their Max VO2 through diligent cardiac rehabilitation, their ultimate results were still well below average.

It has previously been described that normal, healthy subjects have decreased exercise performance in a supine vs upright position. However, due to high venous pressures and the need for systemic venous return to overcome gravity in order to perfuse the lungs, one might hypothesize that Fontan patients would have increased exercise performance in a supine vs upright position. The investigators are interested in studying this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* S/p Fontan palliation > 2 years prior
* Age 8 to 30 years

Exclusion Criteria:

* Pacemaker dependence
* Severe hypoxemia (O2 saturation <80%)
* Recent atrial flutter or other arrhythmias
* Protein losing enteropathy (PLE)
* Severe atrioventricular valve regurgitation
* History of cardiac arrest
* Significant comorbidities (renal failure, asthma, etc).

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Fontan-palliated patients aged 8-30 will be recruited for this study. Eligible patients will be identified from the cardiology and surgery database here. Patients will be contacted by phone and/or formal letter informing them of the study. If their primary cardiologist is not in our group, a courtesy call will be made or letter sent. Age and gender matched healthy controls will be sought as well through local recruitment (schools, university campus, local community postings).
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | 40 minutes
  Watts

SECONDARY OUTCOMES:
Peak Oxygen Volume (Peak VO2) | 40 minutes
  milliliters per kilogram of body weight per minute (ml/kg/min)
Peak Heart Rate | 40 minutes
  beats per minute
Peak Pulmonary Artery Pressure | 40 minutes
  millimeters of mercury (mmHg)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Health Systems, Pediatric Cardiology, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Goldstein BH, Connor CE, Gooding L, Rocchini AP. Relation of systemic venous return, pulmonary vascular resistance, and diastolic dysfunction to exercise capacity in patients with single ventricle receiving fontan palliation. Am J Cardiol. 2010 Apr 15;105(8):1169-75. doi: 10.1016/j.amjcard.2009.12.020. Epub 2010 Feb 20. PMID 20381672